CLINICAL TRIAL: NCT03129100
Title: A Multicenter, Long-Term Extension Study of 104 Weeks, Including a Double-Blind, Placebo-Controlled 40-Week Randomized Withdrawal-Retreatment Period, to Evaluate the Maintenance of Treatment Effect of Ixekizumab (LY2439821) in Patients With Axial Spondyloarthritis
Brief Title: A Long Term Extension Study of Ixekizumab (LY2439821) in Participants With Axial Spondyloarthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 16181; I1F-MC-RHBY (Other: Eli Lilly and Company); 2016-002634-69 (EudraCT Number)
Record Dates: First submitted 2017-04-03; First posted 2017-04-26 (Actual); Results first posted 2021-06-18 (Actual); Last update posted 2022-06-13 (Actual); Status verified 2022-05

CONDITIONS: Axial Spondyloarthritis
MeSH Terms: conditions — Axial Spondyloarthritis | interventions — ixekizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Ixekizumab (IXE) 80Q4W (Experimental): Participants received 80 milligram (mg) of Ixekizumab subcutaneously (SC) every four weeks (Q4W).
  Interventions: Drug: Ixekizumab
- Ixekizumab (IXE) 80Q2W (Experimental): Participants received 80 milligram (mg) of Ixekizumab subcutaneously (SC) every two weeks (Q2W).
  Interventions: Drug: Ixekizumab
- Placebo (Placebo Comparator): Participants received subcutaneous dose of placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ixekizumab — Administered SC
  Other Names: LY2439821
  Arms: Ixekizumab (IXE) 80Q2W; Ixekizumab (IXE) 80Q4W
Drug: Placebo — Administered SC
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate, in participants having achieved a state of sustained remission, if the ixekizumab treatment groups are superior to the placebo group in maintaining response during the randomized withdrawal-retreatment period in participants with axial spondyloarthritis.

ELIGIBILITY:
Inclusion Criteria:

* Have completed the final study visit in Study RHBV (NCT02696785), RHBW (NCT02696798), or RHBX (NCT02757352).

(Note: Participants from Study RHBX are not eligible if they permanently discontinued ixekizumab and were receiving a tumor necrosis factor [TNF] inhibitor).

* Must agree to use a reliable method of birth control.

Exclusion Criteria:

* Have significant uncontrolled disorders or abnormal laboratory values that, in the opinion of the investigator, pose an unacceptable risk to the participant if investigational product continues to be administered.
* Have a known hypersensitivity to ixekizumab or any component of this investigational product.
* Had investigational product permanently discontinued during a previous ixekizumab study.
* Had temporary investigational product interruption at any time during or at the final study visit of a previous ixekizumab study and, in the opinion of the investigator, restarting ixekizumab poses an unacceptable risk for the participant's participation in the study.
* Have any other condition that, in the opinion of the investigator, renders the participant unable to understand the nature, scope, and possible consequences of the study or precludes the participant from following and completing the protocol.
* Are currently enrolled in any other clinical trial involving an investigational product or any other type of medical research judged not to be scientifically or medically compatible with this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 773 (Actual)
Dates: Start 2017-05-09 (Actual); Primary Completion 2020-05-26 (Actual); Study Completion 2021-05-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (127):
- United States (23):
  - Arizona Arthritis & Rheumatology Research, Phoenix, Arizona
  - Care Access Research - Huntington Beach, Huntington Beach, California
  - Desert Medical Advances, Palm Desert, California
  - Arthritis Assoc. & Osteoporosis Ctr of Colorado Springs, LLC, Colorado Springs, Colorado
  - Clinical Research Center of CT/NY, Danbury, Connecticut
  - Arthritis Rheumatic Disease Specialties, Aventura, Florida
  - Sarasota Arthritis Center, Sarasota, Florida
  - Marietta Rheumatology, Marietta, Georgia
  - Institute of Arthritis Research, Idaho Falls, Idaho
  - Center for Arthritis & Osteoporosis, Elizabethtown, Kentucky
  - Klein and Associates MD, PA, Cumberland, Maryland
  - Klein and Associates MD, PA, Hagerstown, Maryland
  - Arthritis Consultants Inc., St Louis, Missouri
  - Glacier View Research Institute, Kalispell, Montana
  - Physician Research Collaboration, LLC, Lincoln, Nebraska
  - Shanahan Rheumatology & Immunotherapy, PLLC, Raleigh, North Carolina
  - Carolina Arthritis Associates, Wilmington, North Carolina
  - Oregon Health and Science University, Portland, Oregon
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Articularis Healthcare Group, INC dba Columbia Arthritis Ctr, Columbia, South Carolina
  - Articularis Healthcare d/b/a/ Low Country Rheumatology, PA, Summerville, South Carolina
  - Univ of Texas Health Science Center - Houston, Houston, Texas
  - Arthritis Northwest PLLC, Spokane, Washington
- Argentina (6):
  - Clinica Adventista de Belgrano, Ciudad de Buenos Aires, Buenos Aires
  - CER Instituto Medico, Quilmes, Buenos Aires
  - Centro de Enfermedades del Higado y Aparato Digestivo, Rosario, Santa Fe Province
  - Centro Medico Privado de Reumatologia, San Miguel de Tucumán, Tucumán Province
  - Consultorios Reumatologicos Pampa, Ciudad Autonoma de Buenos Aire
  - CIR Centro de Investigacions Reumatologicas, San Miguel de Tucumán
- KH der Barmherzigen Schwestern Wien BetriebsGesmbH, Vienna, Austria
- Brazil (7):
  - CMIP - Centro Mineiro de Pesquisa, Juiz de Fora, Minas Gerais
  - EDUMED - Educação em Saúde Ltda., Curitiba, Paraná
  - CCBR Brasil Centro de Analises e Pesquisas Clínicas LTDA, Rio de Janeiro, Rio de Janeiro
  - Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - LMK Serviços Médicos S/S, Porto Alegre, Rio Grande do Sul
  - Cpclin Centro de Pesquisas Clinicas, São Paulo, São Paulo
  - CIP - Centro Internacional de Pesquisa, Goiás
- Canada (4):
  - University of Alberta Hospital, Edmonton, Alberta
  - St. Clare's Mercy Hospital, St. John's, Newfoundland and Labrador
  - Centre de Recherche Musculo-Squelettique, Trois-Rivières, Quebec
  - Group de recherche en maladies osseuses, Québec
- Czechia (5):
  - Revmaclinic, s.r.o, Brno
  - Interni a revmatologicka ambulance, Inrea s.r.o., Ostrava
  - Arthrohelp s.r.o, Pardubice
  - Revmatologicky ustav, Prague
  - MEDICAL PLUS, s.r.o., Uherské Hradiště
- Finland (3):
  - Helsinki University Hospital, HYKS, Helsinki
  - Terveystalo Kamppi, Helsinki
  - Kiljava Medical Research, Hyvinkää
- France (3):
  - Hôpital Trousseau, CHRU de Tours, Chambray-lès-Tours
  - Centre hospitalier universitaire Lapeyronie, Montpellier
  - Nouvel Hôpital Orléans La Source, Orléans
- Germany (4):
  - Rheumazentrum Prof. Neeck, Bad Doberan, Mecklenburg-Vorpommern
  - Rheumazentrum Ruhrgebiet, Herne, North Rhine-Westphalia
  - Charité Universitätsmedizin Berlin, Berlin
  - HRF Hamburger Rheuma Forschungszentrum, Hamburg
- Hungary (2):
  - Revita Reumatologiai Kft., Budapest
  - Vital Medical Center, Veszprém
- Israel (4):
  - Barzilai Medical Center, Ashkelon
  - Rambam Medical Center, Haifa
  - Rabin Medical Center, Petah Tikva
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Arcispedale Santa Maria Nuova Azienda Ospedaliera di Reggio Emilia, Reggio Emilia, Italy
- Japan (12):
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Kagawa University Hospital, Kita-gun, Kagawa-ken
  - Kochi Medical School Hospital, Nankoku, Kochi
  - Kuwana City Medical Center, Kuwana, Mie-ken
  - Sasebo Chuo Hospital, Sasebo, Nagasaki
  - Osaka University Hospital, Suita-shi, Osaka
  - Juntendo University Hospital, Bunkyo-ku, Tokyo
  - St. Lukes International Hospital, Chuo-Ku, Tokyo
  - Japanese Red Cross Okayama Hospital, Okayama
  - Osaka City General Hospital, Osaka
  - Osaka City University Hospital, Osaka
  - Yamagata University Hospital, Yamagata
- Mexico (7):
  - Ctro Inv en Artritis y Osteoporosis SC, Mexicali, Estado de Baja California
  - Unidad de Investigacion en Enfermedades Cronico Degenerative, Guadalajara, Jalisco
  - Clinica en Investigación en Reumatologia y Obesidad S.C., Guadalajara, Jalisco
  - Hospital Universitario de Monterrey, Monterrey, Nuevo León
  - Centro de Alta Especialidad Reumatologia Inv del Potosi SC, San Luis Potosí City, San Luis Potosí
  - Medical Care and Research, S.A. de C.V., Mérida, Yucatán
  - Investigación y Biomedicina de Chihuahua, SC, Chihuahua City
- Netherlands (2):
  - Academisch Medisch Centrum, Amsterdam
  - Antonius Ziekenhuis, Sneek
- Poland (9):
  - NZOZ ZDROWIE Osteo-Medic, Bialystok
  - Szpital Uniwersytecki nr 2 im. dr J. Biziela, Bydgoszcz
  - Centrum Kliniczno-Badawcze, Elblag
  - Centrum Leczenia Osteoporozy Klinika Zdrowej Kosci, Lodz
  - Lecznica MAK-MED, NZOZ, Nadarzyn
  - Prywatna Praktyka Lekarska P. Hrycaj, Poznan
  - Lubelskie Centrum Diagnostyczne, Świdnik
  - Reumatika Centrum Reumatologii, Warsaw
  - Centrum Medyczne AMED, Warsaw
- Puerto Rico (3):
  - GCM Medical Group PSC, San Juan, PR
  - Latin Clinical Trial Center, San Juan, PR
  - Mindful Medical Research, San Juan, PR
- Romania (2):
  - Spitalul Clinic Sf Maria Bucuresti, Bucharest
  - Sp Clinic Judetean de Urgenta Sf.Apostol Andrei Constanta, Constanța
- Russia (6):
  - V.A. Nasonova Research Institute of Rheumatology, Moscow
  - City Clinical Hospital N1, Moscow
  - Ryazan Regional Clinincal Cardiology Dispensary, Ryazan
  - Clinical Rheumatology Hospital # 25, Saint Petersburg
  - Saratov State Medical University, Saratov
  - Clinical Hospital for Emergency Care, Yaroslavl
- South Korea (10):
  - Kyung Hee University Hospital, Seoul, Korea
  - Seoul St. Mary's Hospital, Seoul, Korea
  - Asan Medical Center, Songpa-gu, Seoul
  - Chungnam National University Hospital, Daejeon
  - Seoul National University Hospital, Seoul
  - Hanyang University Medical Center, Seoul
  - Konkuk University Hospital, Seoul
  - Kyunghee University Hospital at Gangdong, Seoul
  - Gangnam Severance Hospital, Seoul
  - Seoul Municipal Boramae Hospital, Seoul
- Spain (3):
  - Centro de Salud Mental Parc Tauli, Sabadell, Barcelona
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Infanta Luisa, Seville
- Taiwan (5):
  - Chang Gung Memorial Hospital - Kaohsiung, Kaohsiung City
  - Chung Shan Medical University Hospital, Taichung
  - China Medical University Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Chi-Mei Medical Center, Yongkang District
- United Kingdom (5):
  - Wythenshawe Hospital, Wythenshawe, Manchester
  - Norfolk and Norwich Hospital, Norwich, Norfolk
  - Haywood Hospital, Stoke-on-Trent, Staffordshire
  - New Cross Hospital, Wolverhampton, West Midlands
  - Solihull Hospital, Solihull, West Midland

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Deodhar A, Poddubnyy D, Rahman P, Ermann J, Tomita T, Bolce R, Leage SL, Kronbergs A, Johnson C, Araujo J, Leung A, van der Heijde D. Long-Term Safety and Efficacy of Ixekizumab in Patients With Axial Spondyloarthritis: 3-year Data From the COAST Program. J Rheumatol. 2023 Aug;50(8):1020-1028. doi: 10.3899/jrheum.221022. Epub 2023 Feb 15. PMID 36792107
- [Derived] Braun J, Kiltz U, Deodhar A, Tomita T, Dougados M, Bolce R, Sandoval D, Lin CY, Walsh J. Efficacy and safety of ixekizumab treatment in patients with axial spondyloarthritis: 2-year results from COAST. RMD Open. 2022 Jul;8(2):e002165. doi: 10.1136/rmdopen-2021-002165. PMID 35853675
- See also: A Long Term Extension Study of Ixekizumab (LY2439821) in Participants With Axial Spondyloarthritis (COAST-Y) — https://trials.lillytrialguide.com/en-US/trial/4AAJNNvqrukMW8Go2I28OI

RESULTS

PARTICIPANT FLOW:
Recruitment Details: * Lead-In (Period 1): 24 weeks (Week 0 to Week 24)
  * Extension Period including Double-Blind, Placebo-Controlled, Randomized Withdrawal-Retreatment (RWR) (Period 2): 40 weeks (Week 24 to Week 64)
  * Long-Term Extension Period (Period 3): 40 weeks (Week 64 to Week 104)
  * Post-Treatment Follow-Up (Period 4): at least 12 weeks and up to 24 weeks after the date of the participant's ETV or last regularly scheduled visit.
Pre-assignment Details: In Period 2, participants who did not achieve sustained remission were assigned to Group A and continued to receive the ixekizumab(IXE) dose regimen that they were receiving during Period 1. Participants who did achieve sustained remission were assigned to Group B (Randomized Withdrawal Extension(RWE) period) and were randomized 2:1 to either continue their IXE dose or to withdraw to placebo. Participants who experienced a flare in group B were retreated with IXE in Retreatment Extension Period.
Groups:
- IXE 80Q4W-Lead-in Period: Participants received 80 milligram (mg) of Ixekizumab subcutaneously (SC) every four weeks (Q4W) for up to week 24.
- IXE80Q2W-Lead-in Period: Participants received 80 mg of Ixekizumab subcutaneously every two weeks (Q2W) for up to week 24.
- IXE80Q4W-Group A Extension Period: Participants continued to receive uninterrupted Ixekizumab 80 mg Q4W subcutaneous dose during the extension period.
- IXE80Q2W-Group A Extension Period: Participants continued to receive uninterrupted Ixekizumab 80 mg Q2W subcutaneous dose during the extension period.
- IXE80Q4W-Group B-Randomized Withdrawal Extension Period: Participants in the Ixekizumab 80 mg Q4W treatment group (Lead-in) were re randomized to receive Ixekizumab 80 mg Q4W subcutaneous dose at Week 24 in the randomized withdrawal extension period.
- IXE80Q2W-Group B-Randomized Withdrawal Extension Period: Participants in the Ixekizumab 80 mg Q2W treatment group (Lead-in) were re randomized to receive subcutaneous dose of Ixekizumab 80 mg Q2W at Week 24 in the randomized withdrawal extension period.
- Placebo-Group B-Randomized Withdrawal Extension Period: Participants were re-randomized to receive subcutaneous dose of placebo at Week 24 in the randomized withdrawal extension period.
- IXE80Q2W/IXE80Q2W-Retreatment Extension Period: Participants in Group B who received Ixekizumab 80 mg Q2W in Period 2 and experienced a flare were retreated with subcutaneous dose of Ixekizumab 80 mg Q2W during the retreatment long-term extension period.
- IXE80Q4W/IXE80Q4W-Retreatment Extension Period: Participants in Group B who received Ixekizumab 80 mg Q4W in Period 2 and experienced a flare were retreated with subcutaneous dose of Ixekizumab 80 mg Q4W during the retreatment long term extension period.
- PBO/IXE80Q2W-Retreatment Extension Period: Participants in Group B who received placebo in Period 2 and experienced a flare were retreated with subcutaneous dose of Ixekizumab 80 mg Q2W during the retreatment long term extension period.
- PBO/IXE80Q4W-Retreatment Extension Period: Participants in Group B who received placebo in Period 2 and experienced a flare were retreated with subcutaneous dose of Ixekizumab 80 mg Q4W during the retreatment long term extension period.
- IXE80Q2W-group A Long-term Extension Period: Participants from "IXE80Q2W group A extension period" continued to receive same treatment that they were receiving at the end of Period 2.
- IXE80Q4W-group A Long-term Extension Period: Participants from "IXE80Q4W group A extension period" continued to receive same treatment that they were receiving at the end of Period 2.
- IXE80Q2W-Group B-Randomized Withdrawal Long-term Extension Period: Participants from "IXE80Q2W-Group B-Randomized Withdrawal Extension Period" continued to receive same treatment that they were receiving at the end of Period 2.
- IXE80Q4W-Group B-Randomized Withdrawal Long-term Extension Period: Participants from "IXE80Q4W-Group B-Randomized Withdrawal Extension Period" continued to receive same treatment that they were receiving at the end of Period 2.
- PBO-Group B-Randomized Withdrawal Long-term Extension Period: Participants from "Placebo-Group B-Randomized Withdrawal Extension Period" continued to receive same treatment that they were receiving at the end of Period 2.
- IXE80Q2W/IXE80Q2W-Retreatment Long-term Extension Period: Participants in Group B who received Ixekizumab 80 mg Q2W in Period 3 and experienced a flare were retreated with subcutaneous dose of Ixekizumab 80 mg Q2W during the retreatment long-term extension period.
- IXE80Q4W/IXE80Q4W-Retreatment Long-term Extension Period: Participants in Group B who received Ixekizumab 80 mg Q4W in Period 3 and experienced a flare were retreated with subcutaneous dose of Ixekizumab 80 mg Q4W during the retreatment long term extension period.
- PBO/IXE80Q2W-Retreatment Long-term Extension Period: Participants in Group B who received placebo in Period 3 and experienced a flare were retreated with subcutaneous dose of Ixekizumab 80 mg Q2W during the retreatment long term extension period.
- PBO/IXE80Q4W-Retreatment Long-term Extension Period: Participants in Group B who received placebo in Period 3 and experienced a flare were retreated with subcutaneous dose of Ixekizumab 80 mg Q4W during the retreatment long term extension period.
- IXE80Q4W-Group A-Escalation Period: Participants in Group A receiving ixekizumab 80 mg Q4W escalated to ixekizumab 80 mg Q2W in Period 3.
- IXE80Q4W-Randomized Withdrawal Escalation Period: Participants in Group B receiving Ixekizumab 80 mg Q4W escalated to ixekizumab 80 mg Q2W.
- PBO-Randomized Withdrawal Escalation Period: Participants in Group B, who received PBO, experienced a flare and retreated with Ixekizumab 80 mg Q4W, escalated to ixekizumab 80 mg Q2W.
- PBO-follow-up Period; IXE80Q4W-follow-up Period; IXE80Q2W-follow-up Period: Participants did not receive any intervention during Follow-up period.
Period: Lead-In Period (Period 1)
Arm/Group | IXE 80Q4W-Lead-in Period | IXE80Q2W-Lead-in Period | IXE80Q4W-Group A Extension Period | IXE80Q2W-Group A Extension Period | IXE80Q4W-Group B-Randomized Withdrawal Extension Period | IXE80Q2W-Group B-Randomized Withdrawal Extension Period | Placebo-Group B-Randomized Withdrawal Extension Period | IXE80Q2W/IXE80Q2W-Retreatment Extension Period | IXE80Q4W/IXE80Q4W-Retreatment Extension Period | PBO/IXE80Q2W-Retreatment Extension Period | PBO/IXE80Q4W-Retreatment Extension Period | IXE80Q2W-group A Long-term Extension Period | IXE80Q4W-group A Long-term Extension Period | IXE80Q2W-Group B-Randomized Withdrawal Long-term Extension Period | IXE80Q4W-Group B-Randomized Withdrawal Long-term Extension Period | PBO-Group B-Randomized Withdrawal Long-term Extension Period | IXE80Q2W/IXE80Q2W-Retreatment Long-term Extension Period | IXE80Q4W/IXE80Q4W-Retreatment Long-term Extension Period | PBO/IXE80Q2W-Retreatment Long-term Extension Period | PBO/IXE80Q4W-Retreatment Long-term Extension Period | IXE80Q4W-Group A-Escalation Period | IXE80Q4W-Randomized Withdrawal Escalation Period | PBO-Randomized Withdrawal Escalation Period | PBO-follow-up Period | IXE80Q4W-follow-up Period | IXE80Q2W-follow-up Period
Started | 350 | 423 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Received at Least One Dose of Study Drug | 348 | 423 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 335 | 406 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 15 | 17 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 2 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 8 | 8 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 3 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Surgery Programmed | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period2 Extension Period (Group A and B)
Arm/Group | IXE 80Q4W-Lead-in Period | IXE80Q2W-Lead-in Period | IXE80Q4W-Group A Extension Period | IXE80Q2W-Group A Extension Period | IXE80Q4W-Group B-Randomized Withdrawal Extension Period | IXE80Q2W-Group B-Randomized Withdrawal Extension Period | Placebo-Group B-Randomized Withdrawal Extension Period | IXE80Q2W/IXE80Q2W-Retreatment Extension Period | IXE80Q4W/IXE80Q4W-Retreatment Extension Period | PBO/IXE80Q2W-Retreatment Extension Period | PBO/IXE80Q4W-Retreatment Extension Period | IXE80Q2W-group A Long-term Extension Period | IXE80Q4W-group A Long-term Extension Period | IXE80Q2W-Group B-Randomized Withdrawal Long-term Extension Period | IXE80Q4W-Group B-Randomized Withdrawal Long-term Extension Period | PBO-Group B-Randomized Withdrawal Long-term Extension Period | IXE80Q2W/IXE80Q2W-Retreatment Long-term Extension Period | IXE80Q4W/IXE80Q4W-Retreatment Long-term Extension Period | PBO/IXE80Q2W-Retreatment Long-term Extension Period | PBO/IXE80Q4W-Retreatment Long-term Extension Period | IXE80Q4W-Group A-Escalation Period | IXE80Q4W-Randomized Withdrawal Escalation Period | PBO-Randomized Withdrawal Escalation Period | PBO-follow-up Period | IXE80Q4W-follow-up Period | IXE80Q2W-follow-up Period
Started | 0 (Only Extension Period participants were included.) | 0 (Only Extension Period participants were included.) | 255 (Participants who entered extension period (Group A).) | 318 (Participants who entered extension period (Group A).) | 48 (Participants who entered extension period (Group B).) | 54 (Participants who entered extension period (Group B).) | 53 (Participants who entered extension period (Group B).) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Received at Least One Dose of Study Drug | 0 | 0 | 255 | 318 | 47 | 54 | 53 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 234 | 312 | 42 | 45 | 32 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 21 | 6 | 6 | 9 | 21 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 2 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 13 | 5 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Experienced Flare | 0 | 0 | 0 | 0 | 5 | 6 | 19 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 2 (Retreatment Extension Period)
Arm/Group | IXE 80Q4W-Lead-in Period | IXE80Q2W-Lead-in Period | IXE80Q4W-Group A Extension Period | IXE80Q2W-Group A Extension Period | IXE80Q4W-Group B-Randomized Withdrawal Extension Period | IXE80Q2W-Group B-Randomized Withdrawal Extension Period | Placebo-Group B-Randomized Withdrawal Extension Period | IXE80Q2W/IXE80Q2W-Retreatment Extension Period | IXE80Q4W/IXE80Q4W-Retreatment Extension Period | PBO/IXE80Q2W-Retreatment Extension Period | PBO/IXE80Q4W-Retreatment Extension Period | IXE80Q2W-group A Long-term Extension Period | IXE80Q4W-group A Long-term Extension Period | IXE80Q2W-Group B-Randomized Withdrawal Long-term Extension Period | IXE80Q4W-Group B-Randomized Withdrawal Long-term Extension Period | PBO-Group B-Randomized Withdrawal Long-term Extension Period | IXE80Q2W/IXE80Q2W-Retreatment Long-term Extension Period | IXE80Q4W/IXE80Q4W-Retreatment Long-term Extension Period | PBO/IXE80Q2W-Retreatment Long-term Extension Period | PBO/IXE80Q4W-Retreatment Long-term Extension Period | IXE80Q4W-Group A-Escalation Period | IXE80Q4W-Randomized Withdrawal Escalation Period | PBO-Randomized Withdrawal Escalation Period | PBO-follow-up Period | IXE80Q4W-follow-up Period | IXE80Q2W-follow-up Period
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 (Participants who experienced flare in Group B Extension period.) | 5 (Participants who experienced flare in Group B Extension period.) | 9 (Participants who experienced flare in Group B Extension period.) | 10 (Participants who experienced flare in Group B Extension period.) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 5 | 8 | 10 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period3-Long-Term Extension Period A & B
Arm/Group | IXE 80Q4W-Lead-in Period | IXE80Q2W-Lead-in Period | IXE80Q4W-Group A Extension Period | IXE80Q2W-Group A Extension Period | IXE80Q4W-Group B-Randomized Withdrawal Extension Period | IXE80Q2W-Group B-Randomized Withdrawal Extension Period | Placebo-Group B-Randomized Withdrawal Extension Period | IXE80Q2W/IXE80Q2W-Retreatment Extension Period | IXE80Q4W/IXE80Q4W-Retreatment Extension Period | PBO/IXE80Q2W-Retreatment Extension Period | PBO/IXE80Q4W-Retreatment Extension Period | IXE80Q2W-group A Long-term Extension Period | IXE80Q4W-group A Long-term Extension Period | IXE80Q2W-Group B-Randomized Withdrawal Long-term Extension Period | IXE80Q4W-Group B-Randomized Withdrawal Long-term Extension Period | PBO-Group B-Randomized Withdrawal Long-term Extension Period | IXE80Q2W/IXE80Q2W-Retreatment Long-term Extension Period | IXE80Q4W/IXE80Q4W-Retreatment Long-term Extension Period | PBO/IXE80Q2W-Retreatment Long-term Extension Period | PBO/IXE80Q4W-Retreatment Long-term Extension Period | IXE80Q4W-Group A-Escalation Period | IXE80Q4W-Randomized Withdrawal Escalation Period | PBO-Randomized Withdrawal Escalation Period | PBO-follow-up Period | IXE80Q4W-follow-up Period | IXE80Q2W-follow-up Period
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 (This period is to report Long-Term Extension Period participants) | 0 (This period is to report Long-Term Extension Period participants) | 0 (This period is to report Long-Term Extension Period participants) | 0 (This period is to report Long-Term Extension Period participants) | 306 (This period is to report Long-Term Extension Period participants) | 177 (This period is to report Long-Term Extension Period participants) | 45 (This period is to report Long-Term Extension Period participants) | 42 (This period is to report Long-Term Extension Period participants) | 30 (This period is to report Long-Term Extension Period participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 287 | 146 | 40 | 37 | 21 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 19 | 31 | 5 | 5 | 9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 12 | 7 | 4 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Escalated to IXE80Q2W | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 24 | 0 | 2 | 8 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 3 (Flare)
Arm/Group | IXE 80Q4W-Lead-in Period | IXE80Q2W-Lead-in Period | IXE80Q4W-Group A Extension Period | IXE80Q2W-Group A Extension Period | IXE80Q4W-Group B-Randomized Withdrawal Extension Period | IXE80Q2W-Group B-Randomized Withdrawal Extension Period | Placebo-Group B-Randomized Withdrawal Extension Period | IXE80Q2W/IXE80Q2W-Retreatment Extension Period | IXE80Q4W/IXE80Q4W-Retreatment Extension Period | PBO/IXE80Q2W-Retreatment Extension Period | PBO/IXE80Q4W-Retreatment Extension Period | IXE80Q2W-group A Long-term Extension Period | IXE80Q4W-group A Long-term Extension Period | IXE80Q2W-Group B-Randomized Withdrawal Long-term Extension Period | IXE80Q4W-Group B-Randomized Withdrawal Long-term Extension Period | PBO-Group B-Randomized Withdrawal Long-term Extension Period | IXE80Q2W/IXE80Q2W-Retreatment Long-term Extension Period | IXE80Q4W/IXE80Q4W-Retreatment Long-term Extension Period | PBO/IXE80Q2W-Retreatment Long-term Extension Period | PBO/IXE80Q4W-Retreatment Long-term Extension Period | IXE80Q4W-Group A-Escalation Period | IXE80Q4W-Randomized Withdrawal Escalation Period | PBO-Randomized Withdrawal Escalation Period | PBO-follow-up Period | IXE80Q4W-follow-up Period | IXE80Q2W-follow-up Period
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 (This period is to report participants who experienced a flare in Period 3.) | 0 (This period is to report participants who experienced a flare in Period 3.) | 0 (This period is to report participants who experienced a flare in Period 3.) | 0 (This period is to report participants who experienced a flare in Period 3.) | 0 (This period is to report participants who experienced a flare in Period 3.) | 6 (This period is to report participants who experienced a flare in Period 3.) | 4 (This period is to report participants who experienced a flare in Period 3.) | 11 (This period is to report participants who experienced a flare in Period 3.) | 15 (This period is to report participants who experienced a flare in Period 3.) | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 2 | 11 | 12 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Escalated to IXE80Q2W | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 3 (Dose Escalation)
Arm/Group | IXE 80Q4W-Lead-in Period | IXE80Q2W-Lead-in Period | IXE80Q4W-Group A Extension Period | IXE80Q2W-Group A Extension Period | IXE80Q4W-Group B-Randomized Withdrawal Extension Period | IXE80Q2W-Group B-Randomized Withdrawal Extension Period | Placebo-Group B-Randomized Withdrawal Extension Period | IXE80Q2W/IXE80Q2W-Retreatment Extension Period | IXE80Q4W/IXE80Q4W-Retreatment Extension Period | PBO/IXE80Q2W-Retreatment Extension Period | PBO/IXE80Q4W-Retreatment Extension Period | IXE80Q2W-group A Long-term Extension Period | IXE80Q4W-group A Long-term Extension Period | IXE80Q2W-Group B-Randomized Withdrawal Long-term Extension Period | IXE80Q4W-Group B-Randomized Withdrawal Long-term Extension Period | PBO-Group B-Randomized Withdrawal Long-term Extension Period | IXE80Q2W/IXE80Q2W-Retreatment Long-term Extension Period | IXE80Q4W/IXE80Q4W-Retreatment Long-term Extension Period | PBO/IXE80Q2W-Retreatment Long-term Extension Period | PBO/IXE80Q4W-Retreatment Long-term Extension Period | IXE80Q4W-Group A-Escalation Period | IXE80Q4W-Randomized Withdrawal Escalation Period | PBO-Randomized Withdrawal Escalation Period | PBO-follow-up Period | IXE80Q4W-follow-up Period | IXE80Q2W-follow-up Period
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 (Participants who are eligible for dose escalations.) | 0 (Participants who are eligible for dose escalations.) | 0 (Participants who are eligible for dose escalations.) | 0 (Participants who are eligible for dose escalations.) | 77 (Participants who are eligible for dose escalations.) | 5 (Participants who are eligible for dose escalations.) | 4 (Participants who are eligible for dose escalations.) | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 73 | 5 | 4 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Period: Period 4 (Post Treatment Follow-up)
Arm/Group | IXE 80Q4W-Lead-in Period | IXE80Q2W-Lead-in Period | IXE80Q4W-Group A Extension Period | IXE80Q2W-Group A Extension Period | IXE80Q4W-Group B-Randomized Withdrawal Extension Period | IXE80Q2W-Group B-Randomized Withdrawal Extension Period | Placebo-Group B-Randomized Withdrawal Extension Period | IXE80Q2W/IXE80Q2W-Retreatment Extension Period | IXE80Q4W/IXE80Q4W-Retreatment Extension Period | PBO/IXE80Q2W-Retreatment Extension Period | PBO/IXE80Q4W-Retreatment Extension Period | IXE80Q2W-group A Long-term Extension Period | IXE80Q4W-group A Long-term Extension Period | IXE80Q2W-Group B-Randomized Withdrawal Long-term Extension Period | IXE80Q4W-Group B-Randomized Withdrawal Long-term Extension Period | PBO-Group B-Randomized Withdrawal Long-term Extension Period | IXE80Q2W/IXE80Q2W-Retreatment Long-term Extension Period | IXE80Q4W/IXE80Q4W-Retreatment Long-term Extension Period | PBO/IXE80Q2W-Retreatment Long-term Extension Period | PBO/IXE80Q4W-Retreatment Long-term Extension Period | IXE80Q4W-Group A-Escalation Period | IXE80Q4W-Randomized Withdrawal Escalation Period | PBO-Randomized Withdrawal Escalation Period | PBO-follow-up Period | IXE80Q4W-follow-up Period | IXE80Q2W-follow-up Period
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 (This period is to report Follow-Up period participants.) | 0 (This period is to report Follow-Up period participants.) | 0 (This period is to report Follow-Up period participants.) | 25 (This period is to report Follow-Up period participants.) | 223 (This period is to report Follow-Up period participants.) | 453 (This period is to report Follow-Up period participants.)
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 22 | 198 | 411
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 25 | 42
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 20 | 37
Not completed — COVID 19 Restrictions | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Not completed — Missed follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: All randomized participants from extension period (period 2).
Groups:
- IXE80Q4W-Group A Extension Period: Participants received 80 mg of Ixekizumab subcutaneously every four weeks (Q4W) for up to week 24.
- IXE80Q2W-Group A Extension Period: Participants received 80 mg of Ixekizumab subcutaneously every two weeks (Q2W) for up to week 24.
- Total: Total of all reporting groups
Arm/Group | IXE80Q4W-Group A Extension Period | IXE80Q2W-Group A Extension Period | IXE80Q4W-Group B-Randomized Withdrawal Extension Period | IXE80Q2W-Group B-Randomized Withdrawal Extension Period | Placebo-Group B-Randomized Withdrawal Extension Period | Total
Number analyzed (Participants) | 255 | 318 | 48 | 54 | 53 | 728
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 240 | 302 | 48 | 53 | 52 | 695
  >=65 years | 15 | 16 | 0 | 1 | 1 | 33
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68 | 95 | 10 | 14 | 15 | 202
  Male | 187 | 223 | 38 | 40 | 38 | 526
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 61 | 86 | 7 | 14 | 11 | 179
  Not Hispanic or Latino | 166 | 204 | 31 | 35 | 39 | 475
  Unknown or Not Reported | 28 | 28 | 10 | 5 | 3 | 74
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 14 | 11 | 2 | 5 | 4 | 36
  Asian | 54 | 50 | 15 | 15 | 13 | 147
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 0 | 0 | 0 | 2
  White | 183 | 247 | 31 | 31 | 35 | 527
  More than one race | 3 | 8 | 0 | 3 | 1 | 15
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  Argentina | 11 | 18 | 1 | 1 | 2 | 33
  Romania | 1 | 3 | 0 | 1 | 0 | 5
  Hungary | 3 | 2 | 1 | 1 | 0 | 7
  United States | 14 | 30 | 1 | 3 | 2 | 50
  Czechia | 37 | 35 | 5 | 4 | 4 | 85
  Japan | 7 | 9 | 1 | 3 | 1 | 21
  United Kingdom | 4 | 6 | 0 | 1 | 0 | 11
  Spain | 5 | 4 | 0 | 1 | 0 | 10
  Russia | 16 | 30 | 6 | 7 | 6 | 65
  Canada | 3 | 2 | 1 | 0 | 2 | 8
  Netherlands | 0 | 2 | 0 | 0 | 0 | 2
  South Korea | 28 | 23 | 10 | 7 | 8 | 76
  Austria | 1 | 1 | 0 | 1 | 0 | 3
  Taiwan | 17 | 16 | 3 | 5 | 2 | 43
  Finland | 0 | 5 | 0 | 1 | 2 | 8
  Brazil | 7 | 16 | 0 | 0 | 0 | 23
  Poland | 50 | 67 | 13 | 7 | 13 | 150
  Italy | 0 | 1 | 0 | 0 | 0 | 1
  Mexico | 40 | 38 | 5 | 11 | 8 | 102
  Israel | 5 | 3 | 0 | 0 | 1 | 9
  France | 4 | 4 | 0 | 0 | 0 | 8
  Germany | 2 | 3 | 1 | 0 | 2 | 8

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who do Not Experience a Flare (Combined Ixekizumab Treatment)
Description: A flare is defined as Ankylosing Spondylitis Disease Activity Score (ASDAS ≥2.1) at 2 consecutive visits, or ASDAS >3.5 at any visit during Period 2.
  ASDAS is a composite index to assess disease activity in AS. The parameters used for the ASDAS (with high sensitivity C-reactive protein (CRP) as acute phase reactant) are total back pain, patient global, peripheral pain/swelling, duration of morning stiffness and CRP in mg/L. The ASDAScrp is calculated with the following equation: 0.121×total back pain+0.110×patient global+0.073×peripheral pain/swelling+0.058×duration of morning stiffness+0.579×Ln(CRP+1). (CRP is in mg/liter, the range of other variables is from 0(normal) to 10(very severe); Ln represents the natural logarithm). Data from five variables combined to yield a score (0.6361 to no defined upper limit), where higher the score worse the disease activity.
Time Frame: Week 64
Population: Participants who achieved a state of sustained remission and were randomized to 40-week double-blind placebo controlled RWR period (Group B). Missing data was imputed using the nonresponder imputation (NRI) method.
Measure: Number; unit: Percentage of participants
Groups:
- Combined IXE: Participants received 80 mg of Ixekizumab subcutaneously every four weeks (Q4W) and every two weeks (Q2W) during the randomized withdrawal extension period.
- Placebo: Participants received placebo subcutaneously during the randomized withdrawal extension period.
Arm/Group | Combined IXE | Placebo
Number analyzed (Participants) | 102 | 53
Percentage of participants | 83.3 | 54.7
Statistical Analysis 1: Comparison: Combined IXE vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 4.35, 95% CI 2-sided [2.03 to 9.35]

2. Secondary Outcome: Percentage of Participants Who do Not Experience a Flare
Description: as for outcome 1
Time Frame: Week 64
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Groups:
- IXE80Q4W: Participants received 80 mg of Ixekizumab subcutaneously every four weeks (Q4W) during the randomized withdrawal extension period.
- IXE80Q2W: Participants received 80 mg of Ixekizumab subcutaneously every two weeks (Q2W) during the randomized withdrawal extension period.
Arm/Group | IXE80Q4W | IXE80Q2W | Placebo
Number analyzed (Participants) | 48 | 54 | 53
Percentage of participants | 83.3 | 83.3 | 54.7
Statistical Analysis 1: Comparison: IXE80Q4W vs Placebo; Test type: Superiority; p = 0.003, Regression, Logistic; Odds Ratio (OR) = 4.28, 95% CI 2-sided [1.66 to 11.03]
Statistical Analysis 2: Comparison: IXE80Q2W vs Placebo; Test type: Superiority; p = 0.001, Regression, Logistic; Odds Ratio (OR) = 4.42, 95% CI 2-sided [1.77 to 11.02]

3. Secondary Outcome: Change From Baseline in Modified Stoke Ankylosing Spondylitis Spinal Score (mSASSS)
Description: The mSASSS is a four-point scoring system for lateral radiographs of the lumbar and cervical spine and has been shown to reliably track disease progression over time, where: 0 = normal; 1 = sclerosis, squaring or erosion; 2 = syndesmophyte; 3 = bony bridge.
  By the scoring system of mSASSS of the spinal x-rays, a total of 24 sites were scored on the lateral cervical and lumbar spine: the anterior corners of the vertebrae from lower border of C2 to upper border T1 (inclusive), and from lower border of T12 to upper border of S1 (inclusive). Each corner was scored from 0 to 3, resulting in a range from 0 [no change] to 72 [progression].
Time Frame: Baseline, 2 Years
Population: Ixekizumab structure population who have been treated with ixekizumab for at least 24 months.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Groups:
- IXE80Q4W: Participants received 80 mg of Ixekizumab subcutaneously every four weeks (Q4W).
- IXE80Q2W: Participants received 80 mg of Ixekizumab subcutaneously every two weeks (Q2W).
- Combined IXE: Participants received 80 mg of Ixekizumab subcutaneously every four weeks (Q4W) and two weeks (Q2W).
Arm/Group | IXE80Q4W | IXE80Q2W | Combined IXE
Number analyzed (Participants) | 115 | 115 | 230
Units on a Scale | 0.41 (2.102) | 0.23 (1.387) | 0.32 (1.779)

4. Secondary Outcome: Percentage of Participants Achieving an Assessment of Spondyloarthritis International Society (ASAS)20 Response
Description: ASAS20 response is defined as a ≥20% improvement and an absolute improvement from baseline of ≥1 units (range 0 to 10) in ≥3 of 4 domains, and no worsening of ≥20% and ≥1 unit (range 0 to 10) in the remaining domain.
  The following ASAS domains are used:
  Patient Global: How active was your spondylitis on average during the last week? score ranges 0 (not active) to 10 (very active).
  Spinal Pain: How much Pain of your spine due to Ankylosing spondylitis? score ranges 0 (no pain) to 10 (severe pain).
  Bath Ankylosing Spondylitis Functional Index (BASFI): Participant asked to rate the difficulty associated with 10 individual basic functional activities. Participant response was captured using Numeric Rating Scale (NRS) (range 0 to 10) with a higher score indicating worse function.
  Inflammation based on mean of Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) Q5 & Q6 (mean of intensity & duration of stiffness): Score ranges from "0" (none) and "10" (very severe).
Time Frame: Week 64
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | IXE80Q4W | IXE80Q2W | Placebo
Number analyzed (Participants) | 48 | 54 | 53
Percentage of participants | 81.3 | 81.5 | 50.9
Statistical Analysis 1: Comparison: IXE80Q4W vs Placebo; Test type: Superiority; p = 0.001, Regression, Logistic; Odds Ratio (OR) = 4.51, 95% CI 2-sided [1.78 to 11.41]
Statistical Analysis 2: Comparison: IXE80Q2W vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 4.61, 95% CI 2-sided [1.88 to 11.31]

5. Secondary Outcome: Percentage of Participants Achieving an ASAS40 Response
Description: ASAS40 is defined as a ≥40% improvement and an absolute improvement from baseline of ≥2 units (range of 0 to 10) in at least 3 of the following 4 domains without any worsening in the remaining domain. The following ASAS domains are used:
  Patient Global: How active was your spondylitis on average during the last week? score ranges 0 (not active) to 10 (very active).
  Spinal Pain: How much Pain of your spine due to Ankylosing spondylitis? score ranges 0 (no pain) to 10 (severe pain).
  Bath Ankylosing Spondylitis Functional Index (BASFI): Participant asked to rate the difficulty associated with 10 individual basic functional activities. Participant response was captured using Numeric Rating Scale (NRS) (range 0 to 10) with a higher score indicating worse function.
  Inflammation based on mean of Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) Q5 & Q6 (mean of intensity & duration of stiffness): Score ranges from "0" (none) and "10" (very severe).
Time Frame: Week 64
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | IXE80Q4W | IXE80Q2W | Placebo
Number analyzed (Participants) | 48 | 54 | 53
Percentage of Participants | 79.2 | 79.6 | 43.4
Statistical Analysis 1: Comparison: IXE80Q4W vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 5.17, 95% CI 2-sided [2.11 to 12.69]
Statistical Analysis 2: Comparison: IXE80Q2W vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 5.23, 95% CI 2-sided [2.20 to 12.47]

6. Secondary Outcome: Percentage of Participants With Change of Ankylosing Spondylitis Disease Activity Score (ASDAS) ≥1.1 Units
Description: ASDAS is a composite index to assess disease activity in AS. The parameters used for the ASDAS (with CRP as acute phase reactant) are total back pain, patient global, peripheral pain/swelling, duration of morning stiffness and CRP in mg/L. The ASDAScrp is calculated with the following equation: 0.121×total back pain+0.110×patient global+0.073×peripheral pain/swelling+0.058×duration of morning stiffness
  +0.579×Ln(CRP+1). (CRP is in mg/liter, the range of other variables is from 0(normal) to 10(very severe); Ln represents the natural logarithm). Data from five variables combined to yield a score (0.6361 to no defined upper limit), where higher the score worse the disease activity.
Time Frame: Week 64
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | IXE80Q4W | IXE80Q2W | Placebo
Number analyzed (Participants) | 48 | 54 | 53
Percentage of participants | 79.2 | 74.1 | 45.3
Statistical Analysis 1: Comparison: IXE80Q4W vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 4.60, 95% CI 2-sided [1.90 to 11.17]
Statistical Analysis 2: Comparison: IXE80Q2W vs Placebo; Test type: Superiority; p = 0.003, Regression, Logistic; Odds Ratio (OR) = 3.55, 95% CI 2-sided [1.56 to 8.09]

7. Secondary Outcome: Percentage of Participants With Inactive Disease on the ASDAS (<1.3 Units)
Description: ASDAS is a composite index to assess disease activity in AS. The parameters used for the ASDAS (with CRP as acute phase reactant) are total back pain, patient global, peripheral pain/swelling, duration of morning stiffness and CRP in mg/L. The ASDAScrp is calculated with the following equation: 0.121×total back pain+0.110×patient global+0.073×peripheral pain/swelling+0.058×duration of morning stiffness+0.579×Ln(CRP+1). (CRP is in mg/liter, the range of other variables is from 0(normal) to 10(very severe); Ln represents the natural logarithm). Data from five variables combined to yield a score (0.6361 to no defined upper limit), where higher the score worse the disease activity.
Time Frame: Week 64
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | IXE80Q4W | IXE80Q2W | Placebo
Number analyzed (Participants) | 48 | 54 | 53
Percentage of participants | 60.4 | 53.7 | 24.5
Statistical Analysis 1: Comparison: IXE80Q4W vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 4.92, 95% CI 2-sided [2.07 to 11.72]
Statistical Analysis 2: Comparison: IXE80Q2W vs Placebo; Test type: Superiority; p = 0.003, Regression, Logistic; Odds Ratio (OR) = 3.61, 95% CI 2-sided [1.57 to 8.32]

8. Secondary Outcome: Change From Baseline in the Individual Components of the ASAS Criteria
Description: Patient Global: How active was your spondylitis on average during the last week? score ranges 0 (not active) to 10 (very active).
  Spinal Pain: How much Pain of your spine due to Ankylosing spondylitis? score ranges 0 (no pain) to 10 (severe pain).
  Bath Ankylosing Spondylitis Functional Index (BASFI): Participant asked to rate the difficulty associated with 10 individual basic functional activities. Participant response was captured using Numeric Rating Scale (NRS) (range 0 to 10) with a higher score indicating worse function. Inflammation based on Q5 & Q6 mean of Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) (mean of intensity & duration of stiffness): Score ranges from "0" (none) and "10" (very severe). LS mean was determined by ANCOVA with treatment, geographic region, originating study, baseline value and Week 24 value as fixed factors.
Time Frame: Baseline, Week 64
Population: Participants who achieved a state of sustained remission and were randomized to 40-week double-blind placebo controlled RWR period (Group B). Missing data was imputed using the modified baseline observation carried forward (mBOCF) method.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | IXE80Q4W | IXE80Q2W | Placebo
Number analyzed (Participants) | 48 | 54 | 53
Units on a scale
  Patient Global | -5.1 (0.38) | -5.0 (0.36) | -3.0 (0.36)
  Spinal Pain | -5.1 (0.39) | -4.8 (0.37) | -3.0 (0.36)
  BASFI | -4.35 (0.316) | -4.19 (0.301) | -2.79 (0.301)
  Inflammation | -5.20 (0.336) | -4.83 (0.319) | -3.03 (0.317)
Statistical Analysis 1: Comparison: IXE80Q4W vs Placebo; Patient Global; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = -2.1, 95% CI 2-sided [-3.1 to -1.1], Standard Error of Mean 0.51
Statistical Analysis 2: Comparison: IXE80Q2W vs Placebo; Patient Global; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = -2.0, 95% CI 2-sided [-2.9 to -1.0], Standard Error of Mean 0.49
Statistical Analysis 3: Comparison: IXE80Q4W vs Placebo; Spinal Pain; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = -2.1, 95% CI 2-sided [-3.1 to -1.0], Standard Error of Mean 0.51
Statistical Analysis 4: Comparison: IXE80Q2W vs Placebo; Spinal Pain; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = -1.8, 95% CI 2-sided [-2.8 to -0.8], Standard Error of Mean 0.49
Statistical Analysis 5: Comparison: IXE80Q4W vs Placebo; BASFI; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = -1.55, 95% CI 2-sided [-2.39 to -0.72], Standard Error of Mean 0.421
Statistical Analysis 6: Comparison: IXE80Q2W vs Placebo; BASFI; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = -1.40, 95% CI 2-sided [-2.20 to -0.59], Standard Error of Mean 0.409
Statistical Analysis 7: Comparison: IXE80Q4W vs Placebo; Inflammation; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = -2.17, 95% CI 2-sided [-3.05 to -1.28], Standard Error of Mean 0.448
Statistical Analysis 8: Comparison: IXE80Q2W vs Placebo; Inflammation; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = -1.80, 95% CI 2-sided [-2.66 to -0.95], Standard Error of Mean 0.433

9. Secondary Outcome: Percentage of Participants Achieving Bath Ankylosing Spondylitis Disease Activity Index 50 (BASDAI50) Response
Description: The BASDAI is a participant-reported assessment consisting of 6 questions that relate to 5 major symptoms relevant to radiographic axial spondyloarthritis (rad-axSpA): 1) Fatigue, 2) Spinal pain, 3) Peripheral arthritis, 4) Enthesitis, 5) Intensity, and 6) Duration of morning stiffness. Participants need to score each item with a score from 0 to 10 (NRS). Total score is obtained from the average of symptom scores ranging 0 (no problem) to 10 (worst problem), with a higher score indicating more severe AS symptom. BASDAI50 represents an improvement of ≥50% of the BASDAI score from baseline.
Time Frame: Week 64
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | IXE80Q4W | IXE80Q2W | Placebo
Number analyzed (Participants) | 48 | 54 | 53
Percentage of participants | 81.3 | 75.9 | 45.3
Statistical Analysis 1: Comparison: IXE80Q4W vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 5.34, 95% CI 2-sided [2.13 to 13.35]
Statistical Analysis 2: Comparison: IXE80Q2W vs Placebo; Test type: Superiority; p = 0.001, Regression, Logistic; Odds Ratio (OR) = 4.07, 95% CI 2-sided [1.75 to 9.45]

10. Secondary Outcome: Change From Baseline in the Measure of High Sensitivity C-Reactive Protein (CRP)
Description: High sensitivity CRP is the measure of acute phase reactant. It was measured with a high sensitivity assay at the central laboratory to help assess the effect of ixekizumab on disease activity. High sensitivity CRP is a sensitive laboratory assay for serum levels of C-Reactive Protein, which is a biomarker of inflammation. LS mean was determined by ANCOVA with treatment, geographic region, originating study, baseline value and Week 24 value as fixed factors.
Time Frame: Baseline, Week 64
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: milligram per liter (mg/L)
Arm/Group | IXE80Q4W | IXE80Q2W | Placebo
Number analyzed (Participants) | 48 | 54 | 53
milligram per liter (mg/L) | -12.952 (1.4666) | -11.074 (1.3861) | -5.094 (1.3696)
Statistical Analysis 1: Comparison: IXE80Q4W vs Placebo; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = -7.858, 95% CI 2-sided [-11.729 to -3.987], Standard Error of Mean 1.9586
Statistical Analysis 2: Comparison: IXE80Q2W vs Placebo; Test type: Superiority; p = 0.002, ANCOVA; LS Mean Difference = -5.979, 95% CI 2-sided [-9.655 to -2.304], Standard Error of Mean 1.8600

11. Secondary Outcome: Change From Baseline in Bath Ankylosing Spondylitis Metrology Index (BASMI)
Description: BASMI is a combined index comprising of the following 5 clinical measurements of spinal mobility in participants with radiographic axial spondyloarthritis (rad-axSpA).
  1. Lateral Spinal Flexion
  2. Tragus-to-wall distance
  3. Lumbar Flexion (modified Schober)
  4. Maximal intermalleolar distance and
  5. Cervical rotation.
  The BASMI linear result is the average of the 5 assessments and ranges from 0 to 10. The higher the BASMI score the more severe the participant's limitation of movement due to their AS. LS mean was determined by ANCOVA with treatment, geographic region, originating study, baseline value and Week 24 value as fixed factors.
Time Frame: Baseline, Week 64
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | IXE80Q4W | IXE80Q2W | Placebo
Number analyzed (Participants) | 48 | 54 | 53
Units on a scale | -0.69 (0.080) | -0.73 (0.075) | -0.50 (0.073)
Statistical Analysis 1: Comparison: IXE80Q4W vs Placebo; Test type: Superiority; p = 0.062, ANCOVA; LS Mean Difference = -0.20, 95% CI 2-sided [-0.40 to 0.01], Standard Error of Mean 0.104
Statistical Analysis 2: Comparison: IXE80Q2W vs Placebo; Test type: Superiority; p = 0.018, ANCOVA; LS Mean Difference = -0.24, 95% CI 2-sided [-0.43 to -0.04], Standard Error of Mean 0.099

12. Secondary Outcome: Change From Baseline in Chest Expansion in Centimeters
Description: Chest expansion is the difference, in centimeter (cm), between the circumference of the chest in maximal inspiration and maximal expiration. While participants have their hands resting on or behind the head, the assessor will measure the chest encircled length by centimeter (cm) at the fourth intercostal level anteriorly. Two tries were recorded. The better measurement (larger difference) of 2 tries (in centimeters) was used for analyses. LS mean was determined by ANCOVA with treatment, geographic region, originating study, baseline value and Week 24 value as fixed factors.
Time Frame: Baseline, Week 64
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: centimeter (cm)
Arm/Group | IXE80Q4W | IXE80Q2W | Placebo
Number analyzed (Participants) | 48 | 54 | 53
centimeter (cm) | 0.77 (0.256) | 0.53 (0.243) | 0.67 (0.236)
Statistical Analysis 1: Comparison: IXE80Q4W vs Placebo; Test type: Superiority; p = 0.757, ANCOVA; LS Mean Difference = 0.10, 95% CI 2-sided [-0.56 to 0.77], Standard Error of Mean 0.335
Statistical Analysis 2: Comparison: IXE80Q2W vs Placebo; Test type: Superiority; p = 0.670, ANCOVA; LS Mean Difference = -0.14, 95% CI 2-sided [-0.77 to 0.50], Standard Error of Mean 0.322

13. Secondary Outcome: Change From Baseline in Occiput to Wall Distance
Description: The participant is to make a maximum effort to touch the head against the wall when standing with heels and back against the wall (occiput). Then the distance from occiput to wall is measured. Two tries will be recorded. The better (smaller) measurement of 2 tries (in centimeters) will be used for analyses. LS mean was determined by ANCOVA with treatment, geographic region, originating study, baseline value and Week 24 value as fixed factors.
Time Frame: Baseline, Week 64
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: cm
Arm/Group | IXE80Q4W | IXE80Q2W | Placebo
Number analyzed (Participants) | 48 | 54 | 53
cm | -0.78 (0.260) | -0.66 (0.239) | -0.38 (0.235)
Statistical Analysis 1: Comparison: IXE80Q4W vs Placebo; Test type: Superiority; p = 0.236, ANCOVA; LS Mean Difference = -0.40, 95% CI 2-sided [-1.07 to 0.27], Standard Error of Mean 0.338
Statistical Analysis 2: Comparison: IXE80Q2W vs Placebo; Test type: Superiority; p = 0.373, ANCOVA; LS Mean Difference = -0.28, 95% CI 2-sided [-0.92 to 0.35], Standard Error of Mean 0.319

14. Secondary Outcome: Change From Baseline in Maastricht Ankylosing Spondylitis Enthesitis Score (MASES)
Description: The MASES is an index used to measure the severity of enthesitis. The MASES assesses 13 sites for enthesitis using a score of "0" for no activity or "1" for activity. Sites assessed include costochondral 1 (right/left), costochondral 7 (right/left), spinal iliaca anterior superior (right/left), crista iliaca (right/left), spina iliaca posterior (right/left), processus spinosus L5, and Achilles tendon proximal insertion (right/left). The MASES is the sum of all site scores (range 0 to 13); higher scores indicate more severe enthesitis. LS mean was determined by ANCOVA with treatment, geographic region, originating study, baseline value and Week 24 value as fixed factors.
Time Frame: Baseline, Week 64
Population: Participants who achieved a state of sustained remission and were randomized to 40-week double-blind placebo controlled RWR period (Group B), and with Baseline MASES score >0. Missing data was imputed using the modified baseline observation carried forward (mBOCF) method.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | IXE80Q4W | IXE80Q2W | Placebo
Number analyzed (Participants) | 29 | 36 | 35
Units on a scale | -3.55 (0.352) | -3.62 (0.315) | -3.48 (0.302)
Statistical Analysis 1: Comparison: IXE80Q4W vs Placebo; Test type: Superiority; p = 0.885, ANCOVA; LS Mean Difference = -0.07, 95% CI 2-sided [-0.98 to 0.85], Standard Error of Mean 0.459
Statistical Analysis 2: Comparison: IXE80Q2W vs Placebo; Test type: Superiority; p = 0.735, ANCOVA; LS Mean Difference = -0.14, 95% CI 2-sided [-0.95 to 0.68], Standard Error of Mean 0.410

15. Secondary Outcome: Change From Baseline in Spondyloarthritis Research Consortium of Canada (SPARCC) Enthesitis Score
Description: The SPARCC enthesitis is an index used to measure the severity of enthesitis. The SPARCC assesses 16 sites for enthesitis using a score of "0" for no activity or "1" for activity. Sites assessed include Medial epicondyle (left/right [L/R]), Lateral epicondyle (L/R), Supraspinatus insertion into greater tuberosity of humerus (L/R), Greater trochanter (L/R), Quadriceps insertion into superior border of patella (L/R), Patellar ligament insertion into inferior pole of patella or tibial tubercle (L/R), Achilles tendon insertion into calcaneum (L/R), and Plantar fascia insertion into calcaneum (L/R). The SPARCC is the sum of all site scores (range 0 to 16). Higher scores indicate more severe enthesitis. LS mean was determined by ANCOVA with treatment, geographic region, originating study, baseline value and Week 24 value as fixed factors.
Time Frame: Baseline, Week 64
Population: Participants who achieved a state of sustained remission and were randomized to 40-week double-blind placebo controlled RWR period (Group B), and with baseline SPARCC score >0. Missing data was imputed using the modified baseline observation carried forward (mBOCF) method.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | IXE80Q4W | IXE80Q2W | Placebo
Number analyzed (Participants) | 22 | 30 | 30
Units on a scale | -3.23 (0.388) | -3.34 (0.338) | -2.71 (0.335)
Statistical Analysis 1: Comparison: IXE80Q4W vs Placebo; Test type: Superiority; p = 0.294, ANCOVA; LS Mean Difference = -0.53, 95% CI 2-sided [-1.53 to 0.47], Standard Error of Mean 0.501
Statistical Analysis 2: Comparison: IXE80Q2W vs Placebo; Test type: Superiority; p = 0.164, ANCOVA; LS Mean Difference = -0.64, 95% CI 2-sided [-1.54 to 0.27], Standard Error of Mean 0.453

16. Secondary Outcome: Change From Baseline in Severity of Peripheral Arthritis by Tender Joint Count (TJC) Score of 46 Joints
Description: The number of tender and painful joints was determined by examination of 46 joints (23 joints on each side of the body). The 46 joints were assessed and classified as tender or not tender. Sum of all joints checked to be tender/painful divided by number of evaluable joints which was multiplied by 46 to obtain TJC score. The scores ranges from 0 (no tender/painful joints) to 46 (all joints tender/painful). LS mean was determined by ANCOVA with treatment, geographic region, originating study, baseline value and Week 24 value as fixed factors.
Time Frame: Baseline, Week 64
Population: Participants who achieved a state of sustained remission and were randomized to 40-week double-blind placebo controlled RWR period (Group B), and with baseline TJC >0. Missing data was imputed using the modified baseline observation carried forward (mBOCF) method.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | IXE80Q4W | IXE80Q2W | Placebo
Number analyzed (Participants) | 27 | 33 | 23
Units on a scale | -6.1 (0.76) | -5.3 (0.74) | -4.0 (0.85)
Statistical Analysis 1: Comparison: IXE80Q4W vs Placebo; Test type: Superiority; p = 0.063, ANCOVA; LS Mean Difference = -2.1, 95% CI 2-sided [-4.3 to 0.1], Standard Error of Mean 1.10
Statistical Analysis 2: Comparison: IXE80Q2W vs Placebo; Test type: Superiority; p = 0.211, ANCOVA; LS Mean Difference = -1.3, 95% CI 2-sided [-3.3 to 0.7], Standard Error of Mean 1.02

17. Secondary Outcome: Change From Baseline in Severity of Peripheral Arthritis by Swollen Joint Count (SJC) Score of 44 Joints
Description: The number of swollen joints was determined by examination of 44 joints (22 joints on each side of the body). The 44 joints were assessed and classified as swollen or not swollen. Sum of all joints checked to be swollen divided by number of evaluable joints which was multiplied by 44 to obtain SJC score. The SJC score ranges from 0 (no swollen joints) to 44 (all joints swollen). LS mean was determined by ANCOVA with treatment, geographic region, originating study, baseline value and Week 24 value as fixed factors.
Time Frame: Baseline, Week 64
Population: Participants who achieved a state of sustained remission and were randomized to 40-week double-blind placebo controlled RWR period (Group B), and with baseline SJC >0. Missing data was imputed using the modified baseline observation carried forward (mBOCF) method.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | IXE80Q4W | IXE80Q2W | Placebo
Number analyzed (Participants) | 16 | 21 | 15
Units on a scale | -3.6 (0.67) | -3.9 (0.59) | -2.7 (0.73)
Statistical Analysis 1: Comparison: IXE80Q4W vs Placebo; Test type: Superiority; p = 0.334, ANCOVA; LS Mean Difference = -0.9, 95% CI 2-sided [-2.7 to 0.9], Standard Error of Mean 0.90
Statistical Analysis 2: Comparison: IXE80Q2W vs Placebo; Test type: Superiority; p = 0.168, ANCOVA; LS Mean Difference = -1.2, 95% CI 2-sided [-3.0 to 0.5], Standard Error of Mean 0.88

18. Secondary Outcome: Percentage of Participants With Anterior Uveitis or Uveitis Flares
Description: Anterior uveitis is an inflammation of the middle layer of the eye. which includes the iris (colored part of the eye) and the adjacent tissue, known as the ciliary body.
Time Frame: Week 64
Population: Participants who achieved a state of sustained remission and were randomized to 40-week double-blind placebo controlled RWR period (Group B), and regardless of history of anterior uveitis.
Measure: Number; unit: Percentage of Participants
Arm/Group | IXE80Q4W | IXE80Q2W | Placebo
Number analyzed (Participants) | 48 | 54 | 53
Percentage of Participants | 4.2 | 5.6 | 5.7

19. Secondary Outcome: Change From Baseline in the Fatigue Numeric Rating Scale (NRS) Score
Description: The fatigue severity NRS is a participant administered single-item 11-point horizontal scale anchored at 0 and 10, with 0 representing "no fatigue" and 10 representing "as bad as you can imagine". Participants rate their fatigue (feeling tired or worn out) by circling the 1 number that describes their worst level of fatigue during the previous 24 hours. LS mean was determined by ANCOVA with treatment, geographic region, originating study, baseline value and Week 24 value as fixed factors.
Time Frame: Baseline, Week 64
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | IXE80Q4W | IXE80Q2W | Placebo
Number analyzed (Participants) | 48 | 54 | 53
units on a scale | -4.2 (0.31) | -4.3 (0.29) | -3.5 (0.28)
Statistical Analysis 1: Comparison: IXE80Q4W vs Placebo; Test type: Superiority; p = 0.100, ANCOVA; LS Mean Difference = -0.7, 95% CI 2-sided [-1.5 to 0.1], Standard Error of Mean 0.40
Statistical Analysis 2: Comparison: IXE80Q2W vs Placebo; Test type: Superiority; p = 0.047, ANCOVA; LS Mean Difference = -0.8, 95% CI 2-sided [-1.5 to -0.0], Standard Error of Mean 0.38

20. Secondary Outcome: Change From Baseline on the Quick Inventory of Depressive Symptomatology Self-Report-16 (QIDS-SR16)
Description: The 16-item QIDS-SR16 version is a widely used validated scale designed to assess the severity of depressive symptoms. The participant was asked to rate the severity and frequency of specific symptoms present over the last 7 days. The QIDS-SR16 total scores range from 0 to 27, where higher scores indicate higher severity of symptoms. LS mean was determined by ANCOVA with treatment, geographic region, originating study, baseline value and Week 24 value as fixed factors.
Time Frame: Baseline, Week 64
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | IXE80Q4W | IXE80Q2W | Placebo
Number analyzed (Participants) | 48 | 54 | 53
units on a scale | -3.68 (0.362) | -3.28 (0.344) | -2.80 (0.342)
Statistical Analysis 1: Comparison: IXE80Q4W vs Placebo; Test type: Superiority; p = 0.068, ANCOVA; LS Mean Difference = -0.88, 95% CI 2-sided [-1.83 to 0.06], Standard Error of Mean 0.479
Statistical Analysis 2: Comparison: IXE80Q2W vs Placebo; Test type: Superiority; p = 0.307, ANCOVA; LS Mean Difference = -0.48, 95% CI 2-sided [-1.40 to 0.44], Standard Error of Mean 0.465

21. Secondary Outcome: Change From Baseline in 36-Item Short Form Health Survey (SF-36) Physical Component Summary (PCS) Score
Description: The SF-36 is a 36-item participant administered measure designed to be a short, multipurpose assessment of health in the areas of physical functioning, role - physical, role - emotional, bodily pain, vitality, social functioning, mental health, and general health. The 2 overarching domains of mental well- being and physical well-being are captured by the Mental Component Summary and Physical Component Summary scores. T-scores are used for analysis. The summary scores range from 0 to 100, with higher scores indicating better levels of function and/or better health. LS mean was determined by ANCOVA with treatment, geographic region, originating study, baseline value and Week 24 value as fixed factors.
Time Frame: Baseline, Week 64
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | IXE80Q4W | IXE80Q2W | Placebo
Number analyzed (Participants) | 48 | 54 | 53
units on a scale | 13.2954 (1.1210) | 13.1030 (1.0457) | 10.6934 (1.0366)
Statistical Analysis 1: Comparison: IXE80Q4W vs Placebo; Test type: Superiority; p = 0.079, ANCOVA; LS Mean Difference = 2.6021, 95% CI 2-sided [-0.3011 to 5.5053], Standard Error of Mean 1.4684
Statistical Analysis 2: Comparison: IXE80Q2W vs Placebo; Test type: Superiority; p = 0.087, ANCOVA; LS Mean Difference = 2.4096, 95% CI 2-sided [-0.3541 to 5.1734], Standard Error of Mean 1.3978

22. Secondary Outcome: Change From Baseline in SF-36 Mental Component Summary (MCS) Score
Description: as for outcome 21
Time Frame: Baseline, Week 64
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | IXE80Q4W | IXE80Q2W | Placebo
Number analyzed (Participants) | 48 | 54 | 53
units on a scale | 3.1766 (0.8968) | 4.6404 (0.8369) | 2.3396 (0.8314)
Statistical Analysis 1: Comparison: IXE80Q4W vs Placebo; Test type: Superiority; p = 0.477, ANCOVA; LS Mean Difference = 0.8370, 95% CI 2-sided [-1.4864 to 3.1605], Standard Error of Mean 1.1752
Statistical Analysis 2: Comparison: IXE80Q2W vs Placebo; Test type: Superiority; p = 0.042, ANCOVA; LS Mean Difference = 2.3009, 95% CI 2-sided [0.0880 to 4.5138], Standard Error of Mean 1.1192

23. Secondary Outcome: Change From Baseline in ASAS Health Index (ASAS HI)
Description: The ASAS Health Index (ASAS HI) is a disease specific health-index instrument designed to assess the impact of interventions for SpA, including axSpA. The 17 item instrument has scores ranging from 0 (good Health) to 17 (poor Health). Each item consists of 1 question that the participant needs to respond to with either "I agree" (score 1) or "I do not agree (score 0)." A score of "1" is given where the item is affirmed, indicating adverse health. All item scores are summed to give a total score or index. LS mean was determined by ANCOVA with treatment, geographic region, originating study, baseline value and Week 24 value as fixed factors.
Time Frame: Baseline, Week 64
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | IXE80Q4W | IXE80Q2W | Placebo
Number analyzed (Participants) | 48 | 54 | 53
units on a scale | -4.64 (0.393) | -4.37 (0.368) | -3.64 (0.370)
Statistical Analysis 1: Comparison: IXE80Q4W vs Placebo; Test type: Superiority; p = 0.058, ANCOVA; LS Mean Difference = -0.99, 95% CI 2-sided [-2.02 to 0.04], Standard Error of Mean 0.520
Statistical Analysis 2: Comparison: IXE80Q2W vs Placebo; Test type: Superiority; p = 0.147, ANCOVA; LS Mean Difference = -0.72, 95% CI 2-sided [-1.71 to 0.26], Standard Error of Mean 0.497

24. Secondary Outcome: Change From Baseline in the European Quality of Life - 5 Dimensions 5 Level (EQ-5D-5L) UK Population-based Index Score
Description: The European Quality of Life - 5 Dimensions 5 Level (EQ-5D-5L) is a standardized measure of health status used to provide a simple, generic measure of health for clinical and economic appraisal. The EQ-5D-5L consists of 2 components: a descriptive system of the respondent's health and a rating of his/her current health state using a 0- to 100-mm visual analog scale (VAS). The descriptive system comprises the following 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. LS mean was determined by ANCOVA with treatment, geographic region, originating study, baseline value and Week 24 value as fixed factors.
Time Frame: Baseline, Week 64
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | IXE80Q4W | IXE80Q2W | Placebo
Number analyzed (Participants) | 48 | 54 | 53
units on a scale | 0.2877 (0.0252) | 0.2847 (0.0235) | 0.2459 (0.0237)
Statistical Analysis 1: Comparison: IXE80Q4W vs Placebo; Test type: Superiority; p = 0.213, ANCOVA; LS Mean Difference = 0.0418, 95% CI 2-sided [-0.0329 to 0.1164], Standard Error of Mean 0.0334
Statistical Analysis 2: Comparison: IXE80Q2W vs Placebo; Test type: Superiority; p = 0.225, ANCOVA; LS Mean Difference = 0.0388, 95% CI 2-sided [-0.0324 to 0.1101], Standard Error of Mean 0.0319

25. Secondary Outcome: Change From Baseline in the Work Productivity Activity Impairment Spondyloarthritis (WPAI-SpA) Scores
Description: The WPAI-SpA consists of 6 questions to determine employment status, hours missed from work because of SpA, hours missed from work for other reasons, hours actually worked, the degree to which SpA affected work productivity while at work, and the degree to which SpA affected activities outside of work. The WPAI-SpA has been validated in the rad-axSpA participant population. Four scores are derived: percentage of absenteeism, percentage of presenteeism (reduced productivity while at work), an overall work impairment score that combines absenteeism and presenteeism, and percentage of impairment in activities performed outside of work. The computed percentage range for each sub-scale was from 0-100, with higher scores indicating greater impairment and less productivity. LS mean was determined by ANCOVA with treatment, geographic region, originating study, baseline value and Week 24 value as fixed factors.
Time Frame: Baseline, Week 64
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | IXE80Q4W | IXE80Q2W | Placebo
Number analyzed (Participants) | 48 | 54 | 53
units on a scale | -43.58 (3.329) | -40.10 (3.115) | -32.96 (3.099)
Statistical Analysis 1: Comparison: IXE80Q4W vs Placebo; Percentage of Activity Impairment; Test type: Superiority; p = 0.017, ANCOVA; LS Mean Difference = -10.62, 95% CI 2-sided [-19.28 to -1.95], Standard Error of Mean 4.383
Statistical Analysis 2: Comparison: IXE80Q2W vs Placebo; Percentage of Activity Impairment; Test type: Superiority; p = 0.091, ANCOVA; LS Mean Difference = -7.14, 95% CI 2-sided [-15.44 to 1.16], Standard Error of Mean 4.199

26. Secondary Outcome: Change From Baseline in the Jenkins Sleep Evaluation Questionnaire (JSEQ)
Description: The Jenkins Sleep Evaluation Questionnaire (JSEQ) is a 4 item scale designed to estimate sleep problems in clinical research. The JSEQ assesses the frequency of sleep disturbance in 4 categories: 1) trouble falling asleep, 2) waking up several times during the night, 3) having trouble staying asleep (including waking up far too early), and 4) waking up after the usual amount of sleep feeling tired and worn out. Participants report the numbers of days they experience each of these problems in the past month on a 6 point Likert Scale ranging from 0 = "no days" to 5 = "22-30 days. The total JSEQ score ranges from 0 to 20, with higher scores indicating greater sleep disturbance. LS mean was determined by ANCOVA with treatment, geographic region, originating study, baseline value and Week 24 value as fixed factors.
Time Frame: Baseline, Week 64
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | IXE80Q4W | IXE80Q2W | Placebo
Number analyzed (Participants) | 48 | 54 | 53
units on a scale | -4.0 (0.50) | -3.8 (0.47) | -3.6 (0.47)
Statistical Analysis 1: Comparison: IXE80Q4W vs Placebo; Test type: Superiority; p = 0.531, ANCOVA; LS Mean Difference = -0.4, 95% CI 2-sided [-1.7 to 0.9], Standard Error of Mean 0.66
Statistical Analysis 2: Comparison: IXE80Q2W vs Placebo; Test type: Superiority; p = 0.743, ANCOVA; LS Mean Difference = -0.2, 95% CI 2-sided [-1.4 to 1.0], Standard Error of Mean 0.62

27. Secondary Outcome: Percentage of Participants With No New Syndesmophyte Formation
Description: Percentage of participants with no new syndesmophyte formation was measured using the average of 2 selected readers of 3 readers.
Time Frame: Week 56
Population: Ixekizumab structure population who have been treated with Ixekizumab for at least 24 months
Measure: Number; unit: Percentage of participants
Arm/Group | IXE80Q4W | IXE80Q2W
Number analyzed (Participants) | 115 | 115
Percentage of participants | 80.9 | 87.8

28. Secondary Outcome: Percentage of Participants With Anti-Ixekizumab Antibodies
Description: A treatment emergent - antidrug antibody (TE-ADA) positive participant is defined as: a) a participant with a >= 4-fold increase over a positive baseline antibody titer; or b) for a negative baseline titer, a participant with an increase from the baseline to a level of >= 1:10. Percentage was calculated based on the number of evaluable participants and was calculated by number of participants with treatment-emergent positive anti-ixekizumab antibodies / number of evaluable participants * 100%.
Time Frame: Baseline, Week 64
Population: All randomized participants from Group B, who received at least one dose of study drug.
Measure: Number; unit: Percentage of participants
Groups:
- IXE80Q2W: Participants received 80 mg of Ixekizumab subcutaneously (SC) every two weeks (Q2W) during the randomized withdrawal extension period.
Arm/Group | IXE80Q4W | IXE80Q2W | Placebo
Number analyzed (Participants) | 43 | 51 | 45
Percentage of participants | 4.7 | 2.0 | 20.0

ADVERSE EVENTS:
Time Frame: Baseline, up to 128 weeks
Description: All randomized participants received at least one dose of study treatment. There are gender specific adverse events, only occurring in male or female participants. The number of participants exposed has been adjusted accordingly.
Arm/Group | IXE 80Q4W-Lead-in Period | IXE80Q2W-Lead-in Period | IXE80Q4W-Group A Extension Period | IXE80Q2W-Group A Extension Period | IXE80Q4W-Group B-Randomized Withdrawal Extension Period | IXE80Q2W-Group B-Randomized Withdrawal Extension Period | Placebo-Group B-Randomized Withdrawal Extension Period | IXE80Q2W/IXE80Q2W-Retreatment Extension Period | IXE80Q4W/IXE80Q4W-Retreatment Extension Period | PBO/IXE80Q2W-Retreatment Extension Period | PBO/IXE80Q4W-Retreatment Extension Period | IXE80Q2W-group A Long-term Extension Period | IXE80Q4W-group A Long-term Extension Period | IXE80Q2W-Group B-Randomized Withdrawal Long-term Extension Period | IXE80Q4W-Group B-Randomized Withdrawal Long-term Extension Period | PBO-Group B-Randomized Withdrawal Long-term Extension Period | IXE80Q2W/IXE80Q2W-Retreatment Long-term Extension Period | IXE80Q4W/IXE80Q4W-Retreatment Long-term Extension Period | PBO/IXE80Q2W-Retreatment Long-term Extension Period | PBO/IXE80Q4W-Retreatment Long-term Extension Period | IXE80Q4W-Group A-Escalation Period | IXE80Q4W-Randomized Withdrawal Escalation Period | PBO-randomized Withdrawal Escalation Period | PBO-follow-up Period | IXE80Q4W-follow-up Period | IXE80Q2W-follow-up Period
All-Cause Mortality (participants affected / at risk) | 0/348 | 0/423 | 2/255 | 0/318 | 0/47 | 0/54 | 0/53 | 0/6 | 0/5 | 0/9 | 0/10 | 0/306 | 0/177 | 0/45 | 0/42 | 0/30 | 0/6 | 0/4 | 0/11 | 0/15 | 0/77 | 0/5 | 0/4 | 0/25 | 1/223 | 0/453
Serious Adverse Events (participants affected / at risk) | 10/348 | 12/423 | 12/255 | 11/318 | 2/47 | 2/54 | 1/53 | 1/6 | 0/5 | 0/9 | 0/10 | 15/306 | 3/177 | 1/45 | 1/42 | 0/30 | 0/6 | 0/4 | 0/11 | 0/15 | 1/77 | 0/5 | 0/4 | 0/25 | 3/223 | 2/453
Other Adverse Events (participants affected / at risk) | 79/348 | 108/423 | 62/255 | 82/318 | 8/47 | 17/54 | 16/53 | 0/6 | 4/5 | 2/9 | 1/10 | 52/306 | 37/177 | 8/45 | 6/42 | 9/30 | 0/6 | 3/4 | 6/11 | 5/15 | 6/77 | 2/5 | 0/4 | 0/25 | 14/223 | 27/453
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | IXE 80Q4W-Lead-in Period (N=348) | IXE80Q2W-Lead-in Period (N=423) | IXE80Q4W-Group A Extension Period (N=255) | IXE80Q2W-Group A Extension Period (N=318) | IXE80Q4W-Group B-Randomized Withdrawal Extension Period (N=47) | IXE80Q2W-Group B-Randomized Withdrawal Extension Period (N=54) | Placebo-Group B-Randomized Withdrawal Extension Period (N=53) | IXE80Q2W/IXE80Q2W-Retreatment Extension Period (N=6) | IXE80Q4W/IXE80Q4W-Retreatment Extension Period (N=5) | PBO/IXE80Q2W-Retreatment Extension Period (N=9) | PBO/IXE80Q4W-Retreatment Extension Period (N=10) | IXE80Q2W-group A Long-term Extension Period (N=306) | IXE80Q4W-group A Long-term Extension Period (N=177) | IXE80Q2W-Group B-Randomized Withdrawal Long-term Extension Period (N=45) | IXE80Q4W-Group B-Randomized Withdrawal Long-term Extension Period (N=42) | PBO-Group B-Randomized Withdrawal Long-term Extension Period (N=30) | IXE80Q2W/IXE80Q2W-Retreatment Long-term Extension Period (N=6) | IXE80Q4W/IXE80Q4W-Retreatment Long-term Extension Period (N=4) | PBO/IXE80Q2W-Retreatment Long-term Extension Period (N=11) | PBO/IXE80Q4W-Retreatment Long-term Extension Period (N=15) | IXE80Q4W-Group A-Escalation Period (N=77) | IXE80Q4W-Randomized Withdrawal Escalation Period (N=5) | PBO-randomized Withdrawal Escalation Period (N=4) | PBO-follow-up Period (N=25) | IXE80Q4W-follow-up Period (N=223) | IXE80Q2W-follow-up Period (N=453)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Iridocyclitis (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis ulcerative (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Crohn's disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Strangulated umbilical hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Soft tissue inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Covid-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Orchitis (Infections and infestations) | 1/256 (1) | 0/293 (0) | 0/187 (0) | 0/223 (0) | 0/37 (0) | 0/40 (0) | 0/38 (0) | 0/4 (0) | 0/4 (0) | 0/7 (0) | 0/8 (0) | 0/215 (0) | 0/130 (0) | 0/34 (0) | 0/33 (0) | 0/21 (0) | 0/4 (0) | 0/3 (0) | 0/8 (0) | 0/12 (0) | 0/56 (0) | 0/3 (0) | 0/1 (0) | 0/17 (0) | 0/166 (0) | 0/317 (0)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Comminuted fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ilium fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal column injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Synovial rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Axial spondyloarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Spinal ligament ossification (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Benign lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/92 (0) | 1/130 (1) | 0/68 (0) | 0/95 (0) | 0/10 (0) | 0/14 (0) | 0/15 (0) | 0/2 (0) | 0/1 (0) | 0/2 (0) | 0/2 (0) | 0/91 (0) | 0/47 (0) | 0/11 (0) | 0/9 (0) | 0/9 (0) | 0/2 (0) | 0/1 (0) | 0/3 (0) | 0/3 (0) | 0/21 (0) | 0/2 (0) | 0/3 (0) | 0/8 (0) | 0/57 (0) | 0/136 (0)
Ovarian germ cell teratoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/92 (0) | 0/130 (0) | 0/68 (0) | 0/95 (0) | 1/10 (1) | 0/14 (0) | 0/15 (0) | 0/2 (0) | 0/1 (0) | 0/2 (0) | 0/2 (0) | 0/91 (0) | 0/47 (0) | 0/11 (0) | 0/9 (0) | 0/9 (0) | 0/2 (0) | 0/1 (0) | 0/3 (0) | 0/3 (0) | 0/21 (0) | 0/2 (0) | 0/3 (0) | 0/8 (0) | 0/57 (0) | 0/136 (0)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral venous sinus thrombosis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemic unconsciousness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myelopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Radiculopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Major depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal colic (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 0/92 (0) | 0/130 (0) | 0/68 (0) | 0/95 (0) | 0/10 (0) | 0/14 (0) | 0/15 (0) | 0/2 (0) | 0/1 (0) | 0/2 (0) | 0/2 (0) | 1/91 (1) | 0/47 (0) | 0/11 (0) | 0/9 (0) | 0/9 (0) | 0/2 (0) | 0/1 (0) | 0/3 (0) | 0/3 (0) | 0/21 (0) | 0/2 (0) | 0/3 (0) | 0/8 (0) | 0/57 (0) | 0/136 (0)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Venous thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Venous thrombosis limb (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | IXE 80Q4W-Lead-in Period (N=348) | IXE80Q2W-Lead-in Period (N=423) | IXE80Q4W-Group A Extension Period (N=255) | IXE80Q2W-Group A Extension Period (N=318) | IXE80Q4W-Group B-Randomized Withdrawal Extension Period (N=47) | IXE80Q2W-Group B-Randomized Withdrawal Extension Period (N=54) | Placebo-Group B-Randomized Withdrawal Extension Period (N=53) | IXE80Q2W/IXE80Q2W-Retreatment Extension Period (N=6) | IXE80Q4W/IXE80Q4W-Retreatment Extension Period (N=5) | PBO/IXE80Q2W-Retreatment Extension Period (N=9) | PBO/IXE80Q4W-Retreatment Extension Period (N=10) | IXE80Q2W-group A Long-term Extension Period (N=306) | IXE80Q4W-group A Long-term Extension Period (N=177) | IXE80Q2W-Group B-Randomized Withdrawal Long-term Extension Period (N=45) | IXE80Q4W-Group B-Randomized Withdrawal Long-term Extension Period (N=42) | PBO-Group B-Randomized Withdrawal Long-term Extension Period (N=30) | IXE80Q2W/IXE80Q2W-Retreatment Long-term Extension Period (N=6) | IXE80Q4W/IXE80Q4W-Retreatment Long-term Extension Period (N=4) | PBO/IXE80Q2W-Retreatment Long-term Extension Period (N=11) | PBO/IXE80Q4W-Retreatment Long-term Extension Period (N=15) | IXE80Q4W-Group A-Escalation Period (N=77) | IXE80Q4W-Randomized Withdrawal Escalation Period (N=5) | PBO-randomized Withdrawal Escalation Period (N=4) | PBO-follow-up Period (N=25) | IXE80Q4W-follow-up Period (N=223) | IXE80Q2W-follow-up Period (N=453)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Iridocyclitis (Eye disorders) | 8 (8) | 5 (5) | 7 (8) | 10 (11) | 2 (2) | 2 (3) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (7) | 6 (6) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 5 (6)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Crohn's disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 3 (4) | 10 (10) | 6 (6) | 5 (6) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Covid-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Gastrointestinal viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 27 (28) | 40 (42) | 27 (33) | 30 (32) | 2 (3) | 4 (6) | 7 (8) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 19 (20) | 17 (19) | 2 (4) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 6 (6)
Pharyngitis (Infections and infestations) | 5 (6) | 9 (10) | 9 (9) | 7 (7) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (7) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 16 (19) | 22 (24) | 7 (7) | 13 (14) | 2 (3) | 4 (4) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 8 (10) | 3 (3) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Vaginal infection (Infections and infestations) | 0/92 (0) | 0/130 (0) | 0/68 (0) | 0/95 (0) | 0/10 (0) | 0/14 (0) | 0/15 (0) | 0/2 (0) | 0/1 (0) | 0/2 (0) | 0/2 (0) | 0/91 (0) | 1/47 (1) | 0/11 (0) | 0/9 (0) | 1/9 (1) | 0/2 (0) | 0/1 (0) | 0/3 (0) | 0/3 (0) | 0/21 (0) | 0/2 (0) | 0/3 (0) | 0/8 (0) | 0/57 (0) | 1/136 (1)
Contusion (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Foreign body in eye (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 (9) | 6 (6) | 5 (7) | 14 (16) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 4 (4) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 5 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 9 (9) | 15 (15) | 3 (3) | 3 (3) | 1 (1) | 3 (3) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Chondrodynia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enthesopathy (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 0/92 (0) | 0/130 (0) | 0/68 (0) | 0/95 (0) | 1/10 (1) | 0/14 (0) | 0/15 (0) | 0/2 (0) | 0/1 (0) | 0/2 (0) | 0/2 (0) | 0/91 (0) | 0/47 (0) | 0/11 (0) | 0/9 (0) | 0/9 (0) | 0/2 (0) | 0/1 (0) | 0/3 (0) | 0/3 (0) | 0/21 (0) | 0/2 (0) | 0/3 (0) | 0/8 (0) | 0/57 (0) | 0/136 (0)
Cold urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (2) | 5 (5) | 1 (1) | 3 (3) | 0 (0) | 1 (3) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Keratomileusis (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2017-06-27): https://cdn.clinicaltrials.gov/large-docs/00/NCT03129100/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-19): https://cdn.clinicaltrials.gov/large-docs/00/NCT03129100/SAP_001.pdf